CLINICAL TRIAL: NCT06093438
Title: Induction Toripalimab and Chemotherapy in Locally Advanced Cervical Cancer Patients With High Risk of Recurrence: A Prospective, Single-Arm, Phase II Trial
Brief Title: Induction Toripalimab and Chemotherapy in Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020230207083952035
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-09

CONDITIONS: Cervical Cancer; Induction Chemotherapy; Immunotherapy
Keywords: cervical cancer; immunotherapy; neoadjuvant chemotherapy; chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction immunotherapy and chemotherapy (Experimental): Patients enrolled in this arm would receive neoadjuvant immunotherapy and chemotherapy before definitive chemoradiation
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Patients enrolled in this arm would receive three cycles of induction treatment before receiving definitive chemoradiotherapy. The specific regimen is: Paclitaxel(135mg/m2,ivd, d1)+cisplatin(75mg/m2,ivd,d1-3)+Toripalimab (240mg,ivd,d1)±bevacizumab(ivd, d1)/q21d. Patients would receive pelvic MRI to evaluate the regression status of tumor after three cycles of induction treatment. Patients with satisfying tumor regression would receive definitive chemoradiotherapy afterwards. During chemoradiotherapy, patients would receive weekly cisplatin (40mg/m2) and 240mg toripalimab every three weeks. After chemoradiotherapy, patients would receive another three cycles of consolidated treatment (regimen identical to induction treatment).

SUMMARY:
To explore the efficacy of incorporating neoadjuvant immunotherapy into neoadjuvant chemotherapy in locally advanced cervical cancer patients with high risk of recurrence.

DETAILED DESCRIPTION:
For locally advanced cervical cancer patients undergoing definitive chemoradiotherapy, distant metastasis has become a major concern. In this study, investigators selected a subgroup of patients with theoretically higher risk of distant metastasis and intensified their systematic treatment by incorporating PD-L1 inhibitors into neoadjuvant chemotherapy, in order to reduce their risk of distant metastasis and achieve good disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated locally advanced cervical cancer patients with clear pathological diagnosis
2. 2019 FIGO stage IIIB-IVA. For patients with stage IIIC disease, the short diameter of their metastatic lymph nodes should ≥1.5cm
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
4. Life expectancy > 6 months
5. Able to tolerate concurrent chemoradiotherapy assessed by researches
6. No obvious active bleeding;
7. Adequate hematological, renal and hepatic functions:
8. No concomitant malignancies
9. Female subjects of childbearing potential should have a negative pregnancy test and must take effective and reliable contraceptive measures during the clinical trial period;
10. Voluntarily-signed informed consent.

Exclusion Criteria:

1. Concomitant other malignancies;
2. Patients with metastatic or recurrent disease;
3. Patients received any form of treatment before enrollment;
4. Severe concomitant chronic diseases (diabetes, hypertension, etc.) or acute infections;
5. Impaired hematological, renal or hepatic functions:

   1. Hemoglobin < 9.0 g/dl
   2. Neutrophils < 2000 cells/μl; Leukocytes < 4 × 109/L
   3. Platelets > 100 × 109/L
   4. Serum ALT/AST > 2.5×UNL
   5. Serum Total bilirubin > 1.5× UNL

   g. Serum urea nitrogen (BUN) > 1.5 × upper normal limit (UNL) h. Serum creatinine (Cr) > 1.5 × upper normal limit (UNL)
6. Patients with obvious arrhythmia, myocardial ischemia, severe atrioventricular block, cardiac insufficiency or severe heart valve disease;
7. Patients with uncontrolled mental diseases;
8. Pregnant or lactating woman;
9. Participating in other clinical trials;
10. Anyone considered not suitable for enrollment by principal investigator;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1
Volume changes of core radiation targets and irradiated normal tissues after induction treatment | 5-year
  Volume change of PTV, PGTVnd, Bladder V45, V50, Dmax, Dmean, Rectum V45, V50, Dmax, Dmean, Bowel bag V45, V50

SECONDARY OUTCOMES:
Progression-free survival | 1-year, 2-year
  Time from diagnosis of disease to disease progression or death due to any cause
Distant metastasis-free survival | 1-year, 2-year
  Time from diagnosis to distant metastasis or death due to any cause
Incidence of treatment-related side effects | 5-year
  Incidence of treatment-related side effects (i.e., radiation-related proctitis, cystitis, ,vaginitis, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Chen, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China